CLINICAL TRIAL: NCT05364801
Title: Impact of Anxiety on the Decision-making Process of Anesthesiologists in the Choice of Drugs for Induction of General Anesthesia of Patients With Aspiration Risk Factors
Brief Title: Impact of Anxiety on the Decision-making Processes of Anesthesiologists
Acronym: DECIDINH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/683
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-10

CONDITIONS: Anxiety; Decision Making; General Anesthesia
MeSH Terms: conditions — Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Online anonymous survey

SUMMARY:
Except for exaggerated situations in which aspiration risk seems obvious (or absent), the choice of a rapid sequence induction protocol for general anesthesia is often made under uncertainty, according to the individual assessment of the balance between the aspiration risk on one hand and the anaphylaxis risk induced by short-acting curares on the other hand.

The impact of anxiety and impulsivity on the choice of induction protocols under uncertainty has never been studied before.

In order to investigate this issue, an online anonymous survey has been designed and will be sent to the anesthesiologists of the Bourgogne Franche-Comté and Grand Est regions in France.

The primary objective of this study is to assess the impact of trait-anxiety using the STAI-Y2 form on the decision-making process of anesthesiologists during the choice of an induction protocol for patients at risk of aspiration.

The secondary objectives are to characterize decision-making profiles, to measure the implicit dimension of anxiety using an Implicit association test, to study the impact of impulsivity on decision-making processes under uncertainty using the short version of UPPS-P scale and to study the role of socio-demographic data and professional history in these decisions.

ELIGIBILITY:
Inclusion Criteria:

* all anesthesiologists who have completed their PhD
* working in France
* in a public or private healthcare facility

Exclusion Criteria:

* residents
* retired anesthesiologists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A first phase will include all anesthesiologists of Bourgogne-Franche-Comté and Grand-Est regions (500 subjects) A second phase will include all anesthesiologists registered in France.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory Form Y2 | at 4 months
  Measure of STAI Y2. A score above the threshold of 49 out of 80 will display a trait-anxiety interfering with the decision-making of the anesthesiologists.

SECONDARY OUTCOMES:
Decision-making profiles | at 4 months
  Characterize decision-making profiles using a survey of 10 clinical situations presenting a variable degree of uncertainty, for which a risk score (RS) has been determined by an expert committee. For each situation, the induction protocol must be chosen among a five-choice list gathered in 3 categories : (1) rapid sequence induction (hypnotic + short-acting curare), (2) short protocol (hypnotic + alfentanil or remifentanil) and (3) standard (hypnotic + sufentanil or remifentanil + cisatracurium). Each category has its own score, so that a protocol score (PS) is attributed to the chosen protocol. Finally, a global score (GS) is calculated for each subject by adding the product of RS x PS of the 10 situations.
  The subjects will be attributed to one of the three profiles according to their global score.
Implicit measure of anxiety | at 4 months
  Measure of the anxiety using the Implicit association test.
Impulsivity measure : (negative) Urgency, (lack of) Premeditation, (lack of) Perseverance, Sensation (seeking) - Positive (urgency) scale (UPPS-P scale) | at 4 months
  Measure of the impulsivity using the short version of the UPPS-P scale which is the (negative) Urgency, (lack of) Premeditation, (lack of) Perseverance, Sensation (seeking) - Positive (urgency) scale.
  This scale measures five dimensions of impulsivity. Each dimension will be scored and compared to the mean and standard deviation of the other profiles and to the mean and standard deviation of the general population.
  A score above the mean of the general population shows a higher tendency to impulsive behaviours in the scored dimension. The higher the scores are, the more impulsive the subjects are.
  Standard values for each dimension :
  Dimensions Mean Standard deviation Negative Urgency 9.38 2.73 Positive Urgency 10.84 2.38 Lack of premeditation 7.98 2.15 Lack of perseverance 7.46 2.41 Sensation seeking 10.55 2.72
Socio-demographics and professional history | at 4 months
  Collection of socio-demographic data : sex, experience, practice in anaesthesic wards where aspiration risk is frequently encountered (digestive OR, emergency OR, obstetrics), region, practice in a public or private facility, time spent on duty (hours per week), coffee and cigarette consumption at work, history of severe anaphylaxis resulting from a rapid sequence induction, history of aspiration resulting from an induction of general anesthesia, emotional issues of severe anaphylaxis or aspiration.

CONTACTS AND LOCATIONS:
Overall Officials: David FERREIRA, PH, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besançon, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: No
The data will be strictly anonymous.

REFERENCES:
- [Background] Stiegler MP, Tung A. Cognitive processes in anesthesiology decision making. Anesthesiology. 2014 Jan;120(1):204-17. doi: 10.1097/ALN.0000000000000073. PMID 24212195
- [Background] Croskerry P. The importance of cognitive errors in diagnosis and strategies to minimize them. Acad Med. 2003 Aug;78(8):775-80. doi: 10.1097/00001888-200308000-00003. PMID 12915363
- [Background] Blumenthal-Barby JS, Krieger H. Cognitive biases and heuristics in medical decision making: a critical review using a systematic search strategy. Med Decis Making. 2015 May;35(4):539-57. doi: 10.1177/0272989X14547740. Epub 2014 Aug 21. PMID 25145577
- [Background] Tversky A, Kahneman D. Judgment under Uncertainty: Heuristics and Biases. Science. 1974 Sep 27;185(4157):1124-31. doi: 10.1126/science.185.4157.1124. PMID 17835457
- [Background] Heine MF, Lake CL. Nature and prevention of errors in anesthesiology. J Surg Oncol. 2004 Dec 1;88(3):143-52. doi: 10.1002/jso.20124. No abstract available. PMID 15562456
- [Background] Croskerry P, Abbass A, Wu AW. Emotional influences in patient safety. J Patient Saf. 2010 Dec;6(4):199-205. doi: 10.1097/pts.0b013e3181f6c01a. PMID 21500605
- [Background] Kozlowski D, Hutchinson M, Hurley J, Rowley J, Sutherland J. The role of emotion in clinical decision making: an integrative literature review. BMC Med Educ. 2017 Dec 15;17(1):255. doi: 10.1186/s12909-017-1089-7. PMID 29246213
- [Background] Heyhoe J, Birks Y, Harrison R, O'Hara JK, Cracknell A, Lawton R. The role of emotion in patient safety: Are we brave enough to scratch beneath the surface? J R Soc Med. 2016 Feb;109(2):52-8. doi: 10.1177/0141076815620614. Epub 2015 Dec 18. PMID 26682568
- [Background] Bommer C, Sullivan S, Campbell K, Ahola Z, Agarwal S, O'Rourke A, Jung HS, Gibson A, Leverson G, Liepert AE. Pre-simulation orientation for medical trainees: An approach to decrease anxiety and improve confidence and performance. Am J Surg. 2018 Feb;215(2):266-271. doi: 10.1016/j.amjsurg.2017.09.038. Epub 2017 Nov 10. PMID 29174166
- [Background] Yerkes RM, Dodson JD. The relation of strength of stimulus to rapidity of habit-formation. J Comp Neurol Psychol. 1908;18(5):459-482.
- [Background] Liu G, Chimowitz H, Isbell LM. Affective influences on clinical reasoning and diagnosis: insights from social psychology and new research opportunities. Diagnosis (Berl). 2022 Jan 4;9(3):295-305. doi: 10.1515/dx-2021-0115. eCollection 2022 Aug 1. PMID 34981701
- [Background] Burgess DJ. Are providers more likely to contribute to healthcare disparities under high levels of cognitive load? How features of the healthcare setting may lead to biases in medical decision making. Med Decis Making. 2010 Mar-Apr;30(2):246-57. doi: 10.1177/0272989X09341751. Epub 2009 Sep 2. PMID 19726783
- [Background] Mosier KL, Fischer UM. Judgment and Decision Making by Individuals and Teams: Issues, Models, and Applications. Rev Hum Factors Ergon. 2010;6(1):198-256.
- [Background] Djulbegovic B, Hozo I, Schwartz A, McMasters KM. Acceptable regret in medical decision making. Med Hypotheses. 1999 Sep;53(3):253-9. doi: 10.1054/mehy.1998.0020. PMID 10580533
- [Background] Allen TJ, Moeller FG, Rhoades HM, Cherek DR. Impulsivity and history of drug dependence. Drug Alcohol Depend. 1998 Apr 1;50(2):137-45. doi: 10.1016/s0376-8716(98)00023-4. PMID 9649965
- [Background] Brady KT, Myrick H, McElroy S. The relationship between substance use disorders, impulse control disorders, and pathological aggression. Am J Addict. 1998 Summer;7(3):221-30. PMID 9702290
- [Background] Herman AM, Critchley HD, Duka T. The role of emotions and physiological arousal in modulating impulsive behaviour. Biol Psychol. 2018 Mar;133:30-43. doi: 10.1016/j.biopsycho.2018.01.014. Epub 2018 Jan 31. PMID 29391179
- [Background] Whiteside SP, Lynam DR. The Five Factor Model and impulsivity: using a structural model of personality to understand impulsivity. Personal Individ Differ. 2001;30(4):669-689.
- [Background] Smyth JM, Wonderlich SA, Heron KE, Sliwinski MJ, Crosby RD, Mitchell JE, Engel SG. Daily and momentary mood and stress are associated with binge eating and vomiting in bulimia nervosa patients in the natural environment. J Consult Clin Psychol. 2007 Aug;75(4):629-38. doi: 10.1037/0022-006X.75.4.629. PMID 17663616
- [Background] Monterosso J, Ainslie G. Beyond discounting: possible experimental models of impulse control. Psychopharmacology (Berl). 1999 Oct;146(4):339-47. doi: 10.1007/pl00005480. PMID 10550485
- [Background] Gray JA. The psychophysiological basis of introversion-extraversion. Behav Res Ther. 1970 Aug;8(3):249-66. doi: 10.1016/0005-7967(70)90069-0. No abstract available. PMID 5470377
- [Background] Gray, J. A. (1981). A critique of Eysenck's theory of personality. In H. J. Eysenck (Ed.). A model for personality (pp. 246-276). Berlin: Springer.
- [Background] Auroy Y, Benhamou D, Pequignot F, Bovet M, Jougla E, Lienhart A. Mortality related to anaesthesia in France: analysis of deaths related to airway complications. Anaesthesia. 2009 Apr;64(4):366-70. doi: 10.1111/j.1365-2044.2008.05792.x. PMID 19317699
- [Background] Warner MA, Meyerhoff KL, Warner ME, Posner KL, Stephens L, Domino KB. Pulmonary Aspiration of Gastric Contents: A Closed Claims Analysis. Anesthesiology. 2021 Aug 1;135(2):284-291. doi: 10.1097/ALN.0000000000003831. PMID 34019629
- [Background] Landreau B, Odin I, Nathan N. [Pulmonary aspiration: epidemiology and risk factors]. Ann Fr Anesth Reanim. 2009 Mar;28(3):206-10. doi: 10.1016/j.annfar.2009.01.020. Epub 2009 Mar 21. French. PMID 19304443
- [Background] Stept WJ, Safar P. Rapid induction-intubation for prevention of gastric-content aspiration. Anesth Analg. 1970 Jul-Aug;49(4):633-6. No abstract available. PMID 5534675
- [Background] Reddy JI, Cooke PJ, van Schalkwyk JM, Hannam JA, Fitzharris P, Mitchell SJ. Anaphylaxis is more common with rocuronium and succinylcholine than with atracurium. Anesthesiology. 2015 Jan;122(1):39-45. doi: 10.1097/ALN.0000000000000512. PMID 25405395
- [Background] Avery P, Morton S, Raitt J, Lossius HM, Lockey D. Rapid sequence induction: where did the consensus go? Scand J Trauma Resusc Emerg Med. 2021 May 13;29(1):64. doi: 10.1186/s13049-021-00883-5. PMID 33985541
- [Background] Klucka J, Kosinova M, Zacharowski K, De Hert S, Kratochvil M, Toukalkova M, Stoudek R, Zelinkova H, Stourac P. Rapid sequence induction: An international survey. Eur J Anaesthesiol. 2020 Jun;37(6):435-442. doi: 10.1097/EJA.0000000000001194. PMID 32221099
- [Background] Sajayan A, Wicker J, Ungureanu N, Mendonca C, Kimani PK. Current practice of rapid sequence induction of anaesthesia in the UK - a national survey. Br J Anaesth. 2016 Sep;117 Suppl 1:i69-i74. doi: 10.1093/bja/aew017. Epub 2016 Feb 24. PMID 26917599
- [Background] Egloff B, Schmukle SC. Predictive validity of an Implicit Association Test for assessing anxiety. J Pers Soc Psychol. 2002 Dec;83(6):1441-55. PMID 12500823
- [Background] Greenwald AG, Farnham SD. Using the implicit association test to measure self-esteem and self-concept. J Pers Soc Psychol. 2000 Dec;79(6):1022-38. doi: 10.1037//0022-3514.79.6.1022. PMID 11138752
- [Background] Carpenter TP, Pogacar R, Pullig C, Kouril M, Aguilar S, LaBouff J, Isenberg N, Chakroff A. Survey-software implicit association tests: A methodological and empirical analysis. Behav Res Methods. 2019 Oct;51(5):2194-2208. doi: 10.3758/s13428-019-01293-3. PMID 31515742
- [Background] Anwyl-Irvine AL, Massonnie J, Flitton A, Kirkham N, Evershed JK. Gorilla in our midst: An online behavioral experiment builder. Behav Res Methods. 2020 Feb;52(1):388-407. doi: 10.3758/s13428-019-01237-x. PMID 31016684
- [Background] Egloff B, Schwerdtfeger A, Schmukle SC. Temporal stability of the implicit association test-anxiety. J Pers Assess. 2005 Feb;84(1):82-8. doi: 10.1207/s15327752jpa8401_14. PMID 15639771
- [Background] de Leeuw JR. jsPsych: a JavaScript library for creating behavioral experiments in a Web browser. Behav Res Methods. 2015 Mar;47(1):1-12. doi: 10.3758/s13428-014-0458-y. PMID 24683129
- [Background] Greenwald AG, Nosek BA, Banaji MR. Understanding and using the implicit association test: I. An improved scoring algorithm. J Pers Soc Psychol. 2003 Aug;85(2):197-216. doi: 10.1037/0022-3514.85.2.197. PMID 12916565
- [Background] Billieux J, Rochat L, Ceschi G, Carre A, Offerlin-Meyer I, Defeldre AC, Khazaal Y, Besche-Richard C, Van der Linden M. Validation of a short French version of the UPPS-P Impulsive Behavior Scale. Compr Psychiatry. 2012 Jul;53(5):609-15. doi: 10.1016/j.comppsych.2011.09.001. Epub 2011 Oct 27. PMID 22036009
- [Background] Auroy Y, Benhamou D, Pequignot F, Jougla E, Lienhart A. [Survey of anaesthesia-related mortality in France: the role of aspiration of gastric contents]. Ann Fr Anesth Reanim. 2009 Mar;28(3):200-5. doi: 10.1016/j.annfar.2008.12.018. Epub 2009 Mar 10. French. PMID 19278807
- [Background] Stiegler MP, Goldhaber-Fiebert SN. Cognitive Errors and Cognitive Aids in Anesthesiology. ASA Newsletter 2013; 77:10-12
- See also: Current guidelines from the French Society of Anaesthesia & Intensive Care Medicine for the airway management in anesthesiology of adults, except for difficult intubation — https://sfar.org/wp-content/uploads/2016/12/2b_AFAR_Texte-Long_.pdf
- See also: Rabault K, Master degree on the subject of the assessment of practice concerning the rapid sequence induction for patient at risk of aspiration in the Poitiers University Hospital — https://www.chu-poitiers.fr/specialites/formation-infirmier-anesthesiste/wp-content/uploads/sites/49/2016/10/Karine-RABAULT-2014.pdf
- See also: C. Schmitz. Workarounds: Manipulating a survey at runtime using Javascript - Implicit association test. Published February 16, 2022. Accessed March 13, 2022 — https://manual.limesurvey.org/index.php?title=Workarounds:_Manipulating_a_survey_at_runtime_using_Javascript&oldid=172243
- See also: Muscle relaxants and reversal in anaesthesia. Guidelines from the French Society of Anaesthesia & Intensive Care Medicine — https://sfar.org/wp-content/uploads/2018/10/2_RFE-CURARE-3.pdf